CLINICAL TRIAL: NCT00289016
Title: A Phase II Study of the Efficacy, Safety and Immunogenicity of OncoVEX^GM-CSF in Patients With Stage IIIc and Stage IV Malignant Melanoma
Brief Title: A Study of Talimogene Laherparepvec in Stage IIIc and Stage IV Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioVex Limited (Industry)
Collaborators: Symbion Research International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002/03
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Results first posted 2015-12-18 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-11

CONDITIONS: Melanoma
Keywords: gene transfer; gene therapy; oncolytic virus; GM-CSF; melanoma
MeSH Terms: conditions — Melanoma | interventions — talimogene laherparepvec

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Talimogene Laherparepvec (Experimental): Participants received talimogene laherparepvec at an initial dose of 10⁶ plaque forming units (PFU)/mL injected into 1 or more tumors with maximum total volume of 4 mL (up to 2 mL per tumor). Subsequent doses of talimogene laherparepvec at 10⁸ PFU/mL began 3 weeks after the first dose and were administered every 2 weeks for up to 15 weeks. After the initial 8 doses, if indications of biological activity were observed, treatment could continue for up to 16 additional doses.
  Interventions: Drug: Talimogene Laherparepvec

INTERVENTIONS:
Drug: Talimogene Laherparepvec — Up to 4 mL of 10⁸ pfu/mL/per intratumoral injection
  Other Names: OncoVEX^GM-CSF; T-VEC; IMLYGIC

SUMMARY:
The primary objective of the study was to assess the clinical efficacy of talimogene laherparepvec in terms of tumor response rates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven stage IIIc (including two or more palpable lymph nodes, extracapsular or in-transit metastases) or stage IV melanoma that is not eligible for curative surgery and who have one or more tumors that are accessible for direct injection.
2. Tumors 0.5 to 10 cm in the longest diameter that are suitable for injection (i.e. not bleeding or weeping).
3. Serum lactate dehydrogenase (LDH) levels ≤ 2.0 times the upper limit of normal.
4. Aged 18 years or more.
5. Eastern Cooperative Oncology Group (ECOG) Performance status 0 or 1.
6. Clinically immunocompetent.
7. Recovered from prior therapy with at least 4 weeks since the last exposure to chemotherapy or radiotherapy.
8. Total white cell count ≥ 3.0 x 10^9/L, platelet count ≥ 80 x 10^9/L.
9. Serum creatinine ≤ 0.2 mmol/L.
10. Bilirubin ≤ 1.5 times the upper limit of the normal range, aspartate aminotransferase (AST)/alanine aminotransferase (ALT) equal to or less than twice the upper limit of the normal range and alkaline phosphatase equal to or less than twice the upper limit of the normal range.

Exclusion Criteria:

1. Participation in any previous melanoma immunotherapy trial within one month prior to entry to this trial or any trial of any other investigational agent within the last month prior to entry to this trial.
2. Tumors to be injected lying in mucosal regions or close to an airway, major blood vessel or spinal cord that, in the opinion of the Investigators, could cause occlusion or compression in the case of tumor swelling or erosion into a major vessel in the case of necrosis.
3. Pregnancy, lactation or lack of effective contraception in women of child-bearing potential; lack of effective contraception in men if the partner is of child-bearing potential; women must have been practising an effective contraceptive method for at least three months prior to entry in to the trial (hormonal contraception or intrauterine device in conjunction with a barrier method OR surgically sterilised). Men must use a condom or be surgically sterilised.
4. Major surgery within the 14 days prior to entry to the trial.
5. Intercurrent serious infections within the 28 days prior to entry to the trial.
6. Life-threatening illness unrelated to cancer.
7. Treatment with antiviral agents within the 14 days prior to entry to the trial.
8. Uncontrolled congestive cardiac failure.
9. Clinically active autoimmune disease.
10. Dermatoses involving or near to the tumors to be injected. Limb tumors may not be injected if active dermatoses are present on the same limb. Trunk and head and neck tumors must not be injected if dermatoses are present within 50 cm of the tumor.
11. Known to test positive for human immunodeficiency virus (HIV), hepatitis B or C or syphilis.
12. Patient only has injectable tumors that are not potentially resectable in the case of tumor necrosis or swelling.
13. Previous history of malignancies of other types that have occurred or recurred within the previous 5 years with the exception of cone biopsied carcinoma of the cervix.
14. Corticosteroid use.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Nemunaitis, MD, Principal Investigator — Mary Crowley Medical Research Center; Rob Coffin, PhD, Study Director — BioVex Limited
Locations (8):
- United States (7):
  - UCSD Cancer Center, Thornton Hospital, La Jolla, California
  - UCLA, Los Angeles, California
  - University of Colorado, Anschutz Cancer Pavillion, Aurora, Colorado
  - Hubert H Humphrey Cancer Center, Robbinsdale, Minnesota
  - Mountainside Hospital, Montclair, New Jersey
  - Columbia University, Department of Surgery, New York, New York
  - Mary Crowely Medical Research Center, Dallas, Texas
- Royal Marsden Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Talimogene Laherparepvec
Started | 50
Completed | 13
Not Completed | 37
Not completed — Disease Progression | 29
Not completed — Death | 2
Not completed — Unrelated Medical Condition or Accident | 2
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 48
  Asian | 1
  Hispanic | 1
Eastern Cooperative Oncology Group (ECOG) Performance [Number; unit: participants] — Scale used to assess how a patient's disease is progressing, how the disease affects the daily living abilities of the patient: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity, ambulatory, able to carry out work of a light nature; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self care, confined to a bed or chair > 50% of waking hours; 4 = Completely disabled, confined to bed or chair; 5 = Dead.
  participants
    0 (Fully active) | 31
    1 (Restrictive but ambulatory) | 19
Tumor, Node, Metastasis (TNM) Disease Stage [Number; unit: participants] — Stage IIIC: Ulcerated lesion and 1 lymph node with macrometastasis; 2-3 nodes with macrometastasis or ≥ 4 metastatic lymph nodes, matted lymph nodes, or in-transit met(s)/satellite(s); Stage IV: M1a: Spread to skin, subcutaneous tissue, or lymph nodes; normal lactate dehydrogenase (LDH) level; M1b: Spread to lungs; normal LDH level; M1c: Spread to all other visceral organs, normal LDH level or any distant disease with elevated LDH level.
  participants
    Stage IIIC | 13
    Stage IVM1a | 13
    Stage IVM1b | 5
    Stage IVM1c | 19

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response Rate
Description: Objective response rate is defined as the percentage of participants with an overall best response of complete response or partial response. The objective response to treatment was assessed by computed tomography (CT) scanning or other clinical measurement using modified Response Evaluation Criteria In Solid Tumors (RECIST). Responses must have been confirmed on two visits not less than 4 weeks apart.
  Tumor burden for a visit was calculated as the sum of the longest diameters of all tumors identified and measured up to that visit. Tumor response at each visit was derived from tumor burden, as follows:
  * Complete response (CR): zero tumor burden
  * Partial response (PR): a 30% or greater decrease in tumor burden
  * Progressive disease (PD): a 20% or greater increase in tumor burden
  * Stable disease (SD): none of the above (a < 30% decrease and < 20% increase in tumor burden)
Time Frame: From enrollment until the data cut-off date of 29 November 2008; Median duration of follow-up was 253 days
Population: Intent-to-treat (ITT) population (all participants who received at least 1 dose of talimogene laherparepvec)
Measure: Number; unit: percentage of participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 50
percentage of participants | 28

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) was calculated from the date of the first talimogene laherparepvec dose to the date of death. Median OS was estimated using the Kaplan-Meier method.
Time Frame: From enrollment until the data cut-off date of 29 November 2008; Median duration of follow-up was 253 days
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 50
days | 448.0 [38 to 1174]

3. Secondary Outcome: Time to Progression
Description: Time to progression was calculated from the date of the first talimogene laherparepvec dose to the first date of documented progressive disease (via clinical symptom or tumor burden assessment) that was not followed by a later response of CR, PR, or stable disease.
  Median time to progression was calculated using the Kaplan-Meier method.
Time Frame: From enrollment until the data cut-off date of 29 November 2008; Median duration of follow-up was 253 days.
Population: ITT population
Measure: Median (Full Range); unit: days
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 50
days | 146.0 [15 to 607]

4. Secondary Outcome: Time to Longest Continuous Response
Description: Time to response was calculated from the date of the first talimogene laherparepvec dose to the initial date of the participant's last response interval.
Time Frame: From enrollment until the data cut-off date of 29 November 2008; Median duration of follow-up was 253 days.
Population: ITT population with an objective response (PR or CR)
Measure: Median (Full Range); unit: days
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 14
days | 100 [72 to 288]

5. Secondary Outcome: Duration of Response
Description: Duration of response was calculated from the initial date of response (CR or PR) until the date of progressive disease (or until last follow up that was CR or PR). Participants could have multiple response periods; in this situation, the last response interval was used for the calculation of duration of response.
Time Frame: From enrollment until the data cut-off date of 29 November 2008; Median duration of follow-up was 253 days.
Population: ITT population with an objective response (PR or CR)
Measure: Median (Full Range); unit: days
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 14
days | 223 [1 to 519]

6. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of an adverse event (AE) was graded according to Common Toxicity Criteria for Adverse Events (CTCAE) Version 3 (1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death).
  Serious adverse events include death, life-threatening events, events requiring or prolonging hospitalization, result in persistent or significant disability/incapacity, or a congenital anomaly/birth defect, or otherwise important medical events that may jeopardise the patient or require intervention to prevent one of the above outcomes.
Time Frame: From first dose of talimogene laherparepvec until 30 days after the last dose; the median (minimum, maximum) duration of treatment was 82 (1, 346) days.
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Talimogene Laherparepvec
Number analyzed (Participants) | 50
participants
  Any adverse event | 48
  Treatment-related adverse event | 39
  Adverse event ≥ grade 3 | 23
  Fatal adverse events | 5
  Serious adverse events | 17
  Discontinued study treatment due to adverse event | 2
  Injection site reactions | 27
  Flu-like symptoms | 42

ADVERSE EVENTS:
Time Frame: The median (minimum, maximum) duration of treatment was 82 (1, 346) days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Talimogene Laherparepvec
Serious Adverse Events (participants affected / at risk) | 17/50
Other Adverse Events (participants affected / at risk) | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=50)
Anaemia (Blood and lymphatic system disorders) | 1
Atrioventricular block complete (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Disease progression (General disorders) | 7
Pyrexia (General disorders) | 2
Pneumonia (Infections and infestations) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Talimogene Laherparepvec (N=50)
Anaemia (Blood and lymphatic system disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal tenderness (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 3
Chest pain (General disorders) | 3
Chills (General disorders) | 23
Fatigue (General disorders) | 16
Influenza like illness (General disorders) | 9
Injection site reaction (General disorders) | 3
Malaise (General disorders) | 3
Oedema peripheral (General disorders) | 3
Pain (General disorders) | 7
Pyrexia (General disorders) | 27
Tenderness (General disorders) | 4
Oral herpes (Infections and infestations) | 3
Blood urea increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 5
Decreased appetite (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 10
Anxiety (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 7
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Skin reaction (Skin and subcutaneous tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.